CLINICAL TRIAL: NCT01794247
Title: Intrathecal Magnesium Associated to Lidocaine Decreases the Incidence of the Transitory Neurologic Syndrome Following Same-day-surgery
Brief Title: Intrathecal Magnesium for Same-day-surgery
Acronym: MAGLIDIT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: low recruitment rate
Sponsor: Hospital General de Ciudad Real (Other)
Collaborators: University of Castilla-La Mancha (Other)
Responsible Party: Principal Investigator, Javier Pascual-Ramirez, MD, PhD, Hospital General de Ciudad Real
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MAGLIDIT-12; 2012-004538-40 (EudraCT Number)
Record Dates: First submitted 2013-02-15; First posted 2013-02-18 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2014-03

CONDITIONS: Transient Neurologic Syndrome
MeSH Terms: interventions — Magnesium Sulfate; Fentanyl; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intrathecal magnesium (Experimental): Intrathecal magnesium sulfate 15% 0,5 mL (75 mg) is added to lidocaine 5% 1 mL (50 mg)as anesthetic adjuvant
  Interventions: Drug: Magnesium sulfate; Drug: Lidocaine
- Intrathecal fentanyl (Active Comparator): Intrathecal fentanyl 0.5 mL (25 micrograms)is added to lidocaine 5% 1 ML (50 mg) as anesthetic adjuvant
  Interventions: Drug: Fentanyl; Drug: Lidocaine

INTERVENTIONS:
Drug: Magnesium sulfate
  Arms: Intrathecal magnesium
Drug: Fentanyl
  Arms: Intrathecal fentanyl
Drug: Lidocaine

SUMMARY:
5% hyperbaric lidocaine has lost its usefulness for same-day-surgery (SDS) anaesthesia because it has been blamed responsible for the so-called transitory neurological syndrome (TNS). This entity appears particularly in patients operated on lithotomy and knee arthroscopy position and obese patients. It is a benign, moderately painful (grade 3-4 out of 10) and self-limited in time, but disturbing enough to be avoided in same-day-surgery cases. Other local anesthetics are not competitive with general anesthesia in time to be discharged home from the SDS unit. The magnesium ion is well-known for its protective properties on cells with electrical activity. The objective is to confirm that the magnesium ion added as adjuvant to intrathecal (IT) lidocaine may antagonize TNS incidence. If this hypothesis could be confirmed, the practical and theoretical consequences would be far-reaching.

The method to achieve our objective would be a double-blinded randomized clinical trial considering two groups of intrathecal lidocaine: with and without added IT magnesium.

ELIGIBILITY:
Inclusion Criteria:

* Same day surgery patients
* Operated in lithotomy or arthroscopy position or obese patients

Exclusion Criteria:

* American Society of Anesthesia 3 or 4 patients
* Younger than 18 or elder than 80 years-old
* Active lumbar pain
* Any short of chronic neurologic disease
* Any short of myopathy
* Pregnant women
* Previous history of allergic or toxic reaction to lidocaine, magnesium or fentanyl

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-04; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Transient Neurologic Syndrome Incidence | 7 postoperative days
  Transitory neurological syndrome appears particularly in patients operated on lithotomy and knee arthroscopy position and obese patients. It is a benign, moderately painful (grade 3-4 out of 10) buttocks-legs pain, self-limited in time, but disturbing enough to be avoided in same-day-surgery cases.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Pascual-Ramírez, Md, PhD, Principal Investigator — Hospital general Universitario de Ciudad Real
Locations (2):
- Spain (2):
  - Hospital General universitario de Ciudad Real, Ciudad Real, Castille-La Mancha
  - Hospital General Universitario de Ciudad Real, Ciudad Real, Ciudad Real

REFERENCES:
- [Background] Jabalameli M, Pakzadmoghadam SH. Adding different doses of intrathecal magnesium sulfate for spinal anesthesia in the cesarean section: A prospective double blind randomized trial. Adv Biomed Res. 2012;1:7. doi: 10.4103/2277-9175.94430. Epub 2012 May 11. PMID 23210066
- [Background] Nath MP, Garg R, Talukdar T, Choudhary D, Chakrabarty A. To evaluate the efficacy of intrathecal magnesium sulphate for hysterectomy under subarachnoid block with bupivacaine and fentanyl: A prospective randomized double blind clinical trial. Saudi J Anaesth. 2012 Jul;6(3):254-8. doi: 10.4103/1658-354X.101217. PMID 23162399
- [Background] Khezri MB, Yaghobi S, Hajikhani M, Asefzadeh S. Comparison of postoperative analgesic effect of intrathecal magnesium and fentanyl added to bupivacaine in patients undergoing lower limb orthopedic surgery. Acta Anaesthesiol Taiwan. 2012 Mar;50(1):19-24. doi: 10.1016/j.aat.2012.03.001. Epub 2012 Mar 31. PMID 22500909
- [Background] Shukla D, Verma A, Agarwal A, Pandey HD, Tyagi C. Comparative study of intrathecal dexmedetomidine with intrathecal magnesium sulfate used as adjuvants to bupivacaine. J Anaesthesiol Clin Pharmacol. 2011 Oct;27(4):495-9. doi: 10.4103/0970-9185.86594. PMID 22096283
- [Background] Khalili G, Janghorbani M, Sajedi P, Ahmadi G. Effects of adjunct intrathecal magnesium sulfate to bupivacaine for spinal anesthesia: a randomized, double-blind trial in patients undergoing lower extremity surgery. J Anesth. 2011 Dec;25(6):892-7. doi: 10.1007/s00540-011-1227-z. Epub 2011 Sep 18. PMID 21928127
- [Background] Mebazaa MS, Ouerghi S, Frikha N, Moncer K, Mestiri T, James MF, Ben Ammar MS. Is magnesium sulfate by the intrathecal route efficient and safe? Ann Fr Anesth Reanim. 2011 Jan;30(1):47-50. doi: 10.1016/j.annfar.2010.12.005. Epub 2011 Jan 13. PMID 21236623
- [Background] Ouerghi S, Fnaeich F, Frikha N, Mestiri T, Merghli A, Mebazaa MS, Kilani T, Ben Ammar MS. The effect of adding intrathecal magnesium sulphate to morphine-fentanyl spinal analgesia after thoracic surgery. A prospective, double-blind, placebo-controlled research study. Ann Fr Anesth Reanim. 2011 Jan;30(1):25-30. doi: 10.1016/j.annfar.2010.10.018. Epub 2010 Dec 8. PMID 21145193
- [Background] Malleeswaran S, Panda N, Mathew P, Bagga R. A randomised study of magnesium sulphate as an adjuvant to intrathecal bupivacaine in patients with mild preeclampsia undergoing caesarean section. Int J Obstet Anesth. 2010 Apr;19(2):161-6. doi: 10.1016/j.ijoa.2009.08.007. Epub 2010 Feb 18. PMID 20171080
- [Background] Ghrab BE, Maatoug M, Kallel N, Khemakhem K, Chaari M, Kolsi K, Karoui A. [Does combination of intrathecal magnesium sulfate and morphine improve postcaesarean section analgesia?]. Ann Fr Anesth Reanim. 2009 May;28(5):454-9. doi: 10.1016/j.annfar.2009.03.004. Epub 2009 May 7. French. PMID 19427159
- [Background] Unlugenc H, Ozalevli M, Gunduz M, Gunasti S, Urunsak IF, Guler T, Isik G. Comparison of intrathecal magnesium, fentanyl, or placebo combined with bupivacaine 0.5% for parturients undergoing elective cesarean delivery. Acta Anaesthesiol Scand. 2009 Mar;53(3):346-53. doi: 10.1111/j.1399-6576.2008.01864.x. Epub 2009 Jan 23. PMID 19173689
- [Background] Jellish WS, Zhang X, Langen KE, Spector MS, Scalfani MT, White FA. Intrathecal magnesium sulfate administration at the time of experimental ischemia improves neurological functioning by reducing acute and delayed loss of motor neurons in the spinal cord. Anesthesiology. 2008 Jan;108(1):78-86. doi: 10.1097/01.anes.0000296109.04010.82. PMID 18156885
- [Background] Arcioni R, Palmisani S, Tigano S, Santorsola C, Sauli V, Romano S, Mercieri M, Masciangelo R, De Blasi RA, Pinto G. Combined intrathecal and epidural magnesium sulfate supplementation of spinal anesthesia to reduce post-operative analgesic requirements: a prospective, randomized, double-blind, controlled trial in patients undergoing major orthopedic surgery. Acta Anaesthesiol Scand. 2007 Apr;51(4):482-9. doi: 10.1111/j.1399-6576.2007.01263.x. PMID 17378788
- [Background] Ozalevli M, Cetin TO, Unlugenc H, Guler T, Isik G. The effect of adding intrathecal magnesium sulphate to bupivacaine-fentanyl spinal anaesthesia. Acta Anaesthesiol Scand. 2005 Nov;49(10):1514-9. doi: 10.1111/j.1399-6576.2005.00793.x. PMID 16223399
- [Background] Buvanendran A, McCarthy RJ, Kroin JS, Leong W, Perry P, Tuman KJ. Intrathecal magnesium prolongs fentanyl analgesia: a prospective, randomized, controlled trial. Anesth Analg. 2002 Sep;95(3):661-6, table of contents. doi: 10.1097/00000539-200209000-00031. PMID 12198056
- [Background] Saeki H, Matsumoto M, Kaneko S, Tsuruta S, Cui YJ, Ohtake K, Ishida K, Sakabe T. Is intrathecal magnesium sulfate safe and protective against ischemic spinal cord injury in rabbits? Anesth Analg. 2004 Dec;99(6):1805-1812. doi: 10.1213/01.ANE.0000138039.04548.3D. PMID 15562076